CLINICAL TRIAL: NCT03038490
Title: The Use of an Oral Mixture of Arginine, Glutamine and Beta-hydroxy-beta-methylbutyrate for the Treatment of Pressure Ulcers
Brief Title: The Use of an Oral Mixture of Arginine, Glutamine and Beta-hydroxy-beta-methylbutyrate for Treatment of Pressure Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Our Lady of Maryknoll Hospital (Other)
Collaborators: Wong Tai Sin Hospital (Unknown)
Responsible Party: Principal Investigator, Lo Kwok Man, Associate Consultant, Our Lady of Maryknoll Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KW/FR-16-167(104-04)
Record Dates: First submitted 2017-01-28; First posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Pressure Ulcers Stage III; Pressure Ulcer, Stage IV
MeSH Terms: conditions — Pressure Ulcer | interventions — Abound vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): The treatment group would be given 2 Sackets of an oral mixture of arginine, glutamine and HMB (ABOUND) every day for a maximum period of 4 weeks, either orally or via enteral feeding.
  Interventions: Dietary Supplement: ABOUND
- Control group (No Intervention): All patients would be assessed by a dietitian to ensure them receiving nutritional support of at least 30 kcal/kg/day and of at least 1.2 g/kg/day of protein regardless of feeding method. During the study period, vitamin C and zinc supplement would not be given.

INTERVENTIONS:
Dietary Supplement: ABOUND — an oral mixture of arginine, glutamine and beta-hydroxy-beta-methylbutyrate
  Arms: Study group

SUMMARY:
To investigate whether an oral nutritional supplement of a mixture of arginine, glutamine and HMB for a maximum period of four weeks is more beneficial than the standard dietary approach to the healing of pressure ulcers, and to examine whether the use of it can reduce admissions and length of hospitalizations for these patients.

DETAILED DESCRIPTION:
All patients would be assessed by a dietitian to ensure them receiving nutritional support of at least 30 kcal/kg/day and of at least 1.2 g/kg/day of protein regardless of feeding method. During the study period, vitamin C and zinc supplement would not be given. Nutritional supplement other than that provided by the dietitian to meet the energy and protein requirement would not be given. The pressure ulcers would be cared according to the "Basic nursing standards for patient care: Wound dressing - Version 5" published by the Hospital Authority Head Office.

The treatment group would also be given 2 Sackets of a mixture of arginine, glutamine and HMB (ABOUND) every day for a maximum period of 4 weeks, either orally or via enteral feeding.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatients of medical and geriatric wards of OLMH and WTSH
2. Aged 18 and older with stage III - IV lesions
3. Patients fed orally or through feeding tubes were included

Exclusion Criteria:

1. Patients with history of using the nutritional supplement (ABOUND) in previous three months
2. Patients with cellulitis, wounds with purulent discharge or osteomyelitis or sepsis
3. Patients requiring protein restriction
4. Patients with poorly controlled diabetes mellitus (latest HbA1C > 8.5) (healing process may be affected
5. Patients under palliative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
percentage change in pressure ulcer area | 4 weeks
change in Pressure Ulcer Scale for Healing (PUSH) | 4 weeks

SECONDARY OUTCOMES:
number of hospital admissions | six months
length of hospitalisation | six months

CONTACTS AND LOCATIONS:
Locations (1):
- Our Lady of Maryknoll Hospital, Wong Tai Sin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cereda E, Gini A, Pedrolli C, Vanotti A. Disease-specific, versus standard, nutritional support for the treatment of pressure ulcers in institutionalized older adults: a randomized controlled trial. J Am Geriatr Soc. 2009 Aug;57(8):1395-402. doi: 10.1111/j.1532-5415.2009.02351.x. Epub 2009 Jun 25. PMID 19563522
- [Background] Wong A, Chew A, Wang CM, Ong L, Zhang SH, Young S. The use of a specialised amino acid mixture for pressure ulcers: a placebo-controlled trial. J Wound Care. 2014 May;23(5):259-60, 262-4, 266-9. doi: 10.12968/jowc.2014.23.5.259. PMID 24810310
- [Background] Cereda E, Klersy C, Serioli M, Crespi A, D'Andrea F; OligoElement Sore Trial Study Group. A nutritional formula enriched with arginine, zinc, and antioxidants for the healing of pressure ulcers: a randomized trial. Ann Intern Med. 2015 Feb 3;162(3):167-74. doi: 10.7326/M14-0696. PMID 25643304